CLINICAL TRIAL: NCT02142049
Title: A Multicenter Study of Ibrutinib and Lenalidomide in Combination With DA-EPOCH-R in Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Ibrutinib and Lenalidomide With Dose Adjusted EPOCH-R in Subjects With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1124-CA
Record Dates: First submitted 2014-05-12; First posted 2014-05-20 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-05

CONDITIONS: Diffuse Large B Cell Lymphoma Relapsed; Diffuse Large B Cell Lymphoma Refractory
Keywords: DLBCL; ABC; GCB; Primary Mediastinal B-cell lymphoma; Pharmacyclics; Lenalidomide; lymphoma; Rituximab; EPOCH; Recommended Phase 2 Dose(RP2D)
MeSH Terms: conditions — Lymphoma | interventions — ibrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: Dose Level 1 (Experimental): Ibrutinib 560 mg PO + DA-EPOCH-R
  Interventions: Drug: Ibrutinib; Drug: DA-EPOCH-R
- Part 1: Dose Level 2 (Experimental): Ibrutinib 560 mg (PO) +lenalidomide 15 mg (PO) + DA-EPOCH-R
  Interventions: Drug: Ibrutinib; Drug: DA-EPOCH-R; Drug: Lenalidomide
- Part 1: Dose Level 3 (Experimental): Ibrutinib 560 mg (PO) +lenalidomide 20 mg (PO) + DA-EPOCH-R
  Interventions: Drug: Ibrutinib; Drug: DA-EPOCH-R; Drug: Lenalidomide
- Part 1: Dose Level 4 (Experimental): Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  Interventions: Drug: Ibrutinib; Drug: DA-EPOCH-R; Drug: Lenalidomide
- Part 2: RP2D (Experimental): Recommended Phase 2 Dose(RP2D): Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  Interventions: Drug: Ibrutinib; Drug: DA-EPOCH-R; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib
Drug: DA-EPOCH-R — Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
Drug: Lenalidomide — Lenalidomide
  Arms: Part 1: Dose Level 2; Part 1: Dose Level 3; Part 1: Dose Level 4; Part 2: RP2D

SUMMARY:
This is a Phase 1b/2, open-label, non-randomized multicenter study to assess the safety and efficacy of ibrutinib and lenalidomide in combination with DA-EPOCH-R in subjects with relapsed/refractory Diffuse Large B-cell Lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, non-randomized multicenter study conducted in 2 parts. Part 1, will determine the MTD of the combination of ibrutinib, lenalidomide and DA-EPOCH-R in subjects with DLBCL.

Ibrutinib will be administered at a fixed dose of 560 mg and lenalidomide will be dose-escalated. DA-EPOCH-R will be given at standard doses.

For Part 2, the MTD determined in Part 1 will be the dose used for all subjects. If no MTD is identified, then subjects in Part 2 will be treated with the maximum administered doses (MAD, treatment doses from dose Level 4).

The primary objective for Part 2 is to determine the ORR of ibrutinib and lenalidomide in combination with DA-EPOCH-R in subjects with ABC DLBCL as analyzed by gene expression profiling when treated at recommended phase 2 dose (RP2D).

ELIGIBILITY:
Major inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Pathologically confirmed relapsed/refractory DLBCL
* Subjects must have ≥1 measurable disease site on CT scan (≥ 1.5 cm in longest dimension).
* Adequate hepatic and renal function:

  * AST or ALT ≤2.5 x ULN
  * Serum Creatinine ≤ 2.0 mg/dL and creatinine clearance ≥60 mL/min/1.73
  * Bilirubin ≤1.5 x ULN
* Adequate hematologic function:

  * ANC >1,000 cells/mm3
  * Platelets ≥75,000 cells/mm3
  * Hemoglobin ≥8.0 g/dL
  * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) must be ≤1.5 x the upper limit of the normal range (ULN)
* Must be registered into the Revlimid REMS™program and be willing to comply with the requirements of Revlimid REMS™.

Major Exclusion Criteria:

* Known central nervous system lymphoma
* Any chemotherapy, external beam radiation therapy, or anti-cancer antibodies within 2 weeks
* Radio- or toxin-immunoconjugates within 10 weeks
* Prior allogenetic stem cell (or other organ) transplant within 6 months or any evidence of active graft-versus-host disease or requirement for immunosuppressants within 28 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Neuenburg, MD, Study Director — Pharmacyclics LLC.
Locations (10):
- United States (10):
  - SITE-1, Duarte, California
  - SITE-2, Los Angeles, California
  - SITE-10, Orange, California
  - SITE-3, Chicago, Illinois
  - SITE-5, Baltimore, Maryland
  - SITE-6, Bethesda, Maryland
  - SITE-4, Ann Arbor, Michigan
  - SITE-8, Albuquerque, New Mexico
  - SITE-9, Stony Brook, New York
  - SITE-7, Charleston, South Carolina

REFERENCES:
- [Derived] Wilson WH, Phillips T, Popplewell L, de Vos S, Chhabra S, Kimball AS, Beaupre D, Huang DW, Wright G, Kwei K, Ping J, Neuenburg JK, Staudt LM. Phase 1b/2 study of ibrutinib and lenalidomide with dose-adjusted EPOCH-R in patients with relapsed/refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2021 Sep;62(9):2094-2106. doi: 10.1080/10428194.2021.1907371. Epub 2021 Apr 15. PMID 33856277

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2: RP2D: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
Period: Overall Study
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1: Dose Level 3 | Part 1: Dose Level 4 | Part 2: RP2D
Started | 3 | 3 | 3 | 6 | 20
Completed | 3 | 3 | 3 | 6 | 20
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1: Dose Level 3 | Part 1: Dose Level 4 | Part 2: RP2D | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 20 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 6 | 11 | 22
  >=65 years | 2 | 0 | 2 | 0 | 9 | 13
Age, Continuous [Median (Full Range); unit: years] | 69 [54 to 89] | 58 [41 to 61] | 67 [58 to 68] | 55 [38 to 61] | 59 [28 to 79] | 58 [28 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 7 | 9
  Male | 3 | 2 | 3 | 5 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 2 | 2
  White | 3 | 2 | 3 | 6 | 15 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 20 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities as a Measure of Safety and Tolerability
Description: Part-1: To determine the maximum tolerated dose (MTD) of the combination of ibrutinib and lenalidomide with dose adjusted EPOCH-R
Time Frame: 1 year after last subjects received the first dose
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: All Treated: Ibrutinib 560 mg (PO) +lenalidomide 0,15, 20, and 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1: Dose Level 3 | Part 1: Dose Level 4 | Part 1: All Treated
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Participants | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With Complete Responses (CR) and Partial Responses (PR) as a Measure of Efficacy-ORR
Description: Part 2 - Overall Response rate will be defined as the proportion of subjects who achieve either a Complete Response or a Partial Response according to the international Working Group Response Criteria for NHL as assessed by investigator.
Time Frame: 1 year after last subjects received the first dose
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Treated at RP2D: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
- ABC Subjects Treated at RP2D: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
  Note: There are only 17 samples available for DLBCL subtype test per GEP. Among of them 14 subjects were identified with ABC.
Arm/Group | All Subjects Treated at RP2D | ABC Subjects Treated at RP2D
Number analyzed (Participants) | 26 | 14
Participants | 16 | 9

3. Secondary Outcome: Number of Participants With Complete Responses (CR) and Partial Responses (PR) as a Measure of Efficacy
Description: Part-1: Overall Response rate (ORR) will defined as the proportion of subjects who achieve either a CR or a PR according to the international Working Group Response Criteria for NHL as assessed by investigator.
Time Frame: 1 year after last subjects received the first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1: Dose Level 3 | Part 1: Dose Level 4 | Part 1: All Treated
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Participants | 1 | 2 | 0 | 3 | 6

4. Secondary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability
Description: Part 2: The frequency (number and percentage) of treatment-emergent adverse events will be reported.
Time Frame: 1 year after last subjects received the first dose
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects Treated at RP2D | ABC Subjects Treated at RP2D
Number analyzed (Participants) | 26 | 14
Participants | 26 | 14

5. Secondary Outcome: Progression Free Survival (PFS) and Overall Survival (OS) as a Measure of Efficacy
Description: Part 2: PFS will be measured as time from first study drug administration to disease progression or death from any cause. OS will be measured from the time of first study drug administration until the date of death using Kaplan-Meier methodology.
Time Frame: From initial dose date until the date of first documented progression or death from any cause, whichever came first, assessed up to approximately 1 year after the last subject received the first dose, up to 36 months at the most.
Measure: Median (Full Range); unit: Months
Groups:
- ABC Subjects Treated at RP2D: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
  Note: There are only 17 samples available for DLBCL subtype test per GEP. Among them 14 subjects were identified with ABC.
Arm/Group | All Subjects Treated at RP2D | ABC Subjects Treated at RP2D
Number analyzed (Participants) | 26 | 14
Months
  Progression Free Survival (PFS) | 4.86 [0.03 to 12.45] | 4.86 [0.03 to 9.69]
  Overall Survival (OS) | 15.84 [0.26 to 28.22] | 15.84 [0.26 to 28.22]

6. Secondary Outcome: Duration of Response (DOR)
Description: Part 2: DOR will be measured from the time by which the measurement criteria are met for CR or PR until the first date by which recurrent or progressive disease is objectively documented.
Time Frame: From initial response date until the date of first documented progression or death from any cause, whichever came first, assessed up to approximately 1 year after the last subject received the first dose.
Measure: Median (Full Range); unit: Months
Groups:
- All Subjects Treated at RP2D Who Achieved Overall Response: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
- ABC Subjects Treated at RP2D Who Achieved Overall Response: Ibrutinib 560 mg (PO) +lenalidomide 25 mg (PO) + DA-EPOCH-R
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
  Note: There are only 17 samples available for DLBCL subtype test per GEP. Among of them 14 subjects were identified with ABC.
Arm/Group | All Subjects Treated at RP2D Who Achieved Overall Response | ABC Subjects Treated at RP2D Who Achieved Overall Response
Number analyzed (Participants) | 16 | 9
Months | 3.94 [0.03 to 10.48] | 4.09 [0.03 to 7.69]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Part 1: Dose Level 1: Ibrutinib 560 mg PO + DA-EPOCH-R + lenalidomide 0 (PO)
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
- Part 1: Dose Level 2: Ibrutinib 560 mg PO + DA-EPOCH-R + lenalidomide 15 (PO)
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
- Part 1: Dose Level 3: Ibrutinib 560 mg PO + DA-EPOCH-R + lenalidomide 20 (PO)
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
- Part 1: Dose Level 4: Ibrutinib 560 mg PO + DA-EPOCH-R + lenalidomide 25 mg (PO)
  DA-EPOCH-R: Etoposide, Prednisone, Doxorubicin, Cyclophosphamide, Vincristine, Rituximab, Pegfilgrastim
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1: Dose Level 3 | Part 1: Dose Level 4 | All Subjects Treated at RP2D
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/6 | 3/26
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/6 | 19/26
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Level 1 (N=3) | Part 1: Dose Level 2 (N=3) | Part 1: Dose Level 3 (N=3) | Part 1: Dose Level 4 (N=6) | All Subjects Treated at RP2D (N=26)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Level 1 (N=3) | Part 1: Dose Level 2 (N=3) | Part 1: Dose Level 3 (N=3) | Part 1: Dose Level 4 (N=6) | All Subjects Treated at RP2D (N=26)
Anaemia (Blood and lymphatic system disorders) | 3 (11) | 3 (29) | 2 (22) | 4 (16) | 12 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (12) | 1 (4) | 1 (7) | 3 (6) | 12 (28)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 1 (5) | 2 (5) | 4 (11)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 1 (1) | 2 (6) | 1 (1) | 6 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (13) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (9) | 1 (3) | 3 (3) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (4) | 3 (10) | 1 (6) | 5 (7) | 12 (21)
Constipation (Gastrointestinal disorders) | 1 (3) | 3 (11) | 2 (4) | 3 (5) | 11 (17)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (8) | 5 (9) | 15 (24)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (3) | 2 (5) | 4 (7)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (2) | 1 (2) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (9)
Fatigue (General disorders) | 2 (3) | 3 (17) | 1 (5) | 5 (6) | 13 (16)
Oedema peripheral (General disorders) | 1 (1) | 3 (8) | 3 (4) | 2 (3) | 7 (8)
Pyrexia (General disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 5 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 3 (4)
Pain (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (5)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (3) | 2 (8) | 1 (2) | 1 (1) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (19) | 1 (6) | 1 (2) | 4 (6)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Immunoglobulins decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (7) | 2 (7) | 2 (20) | 11 (42)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 2 (3) | 1 (3) | 2 (3) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 3 (3) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (8) | 1 (2) | 3 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (7) | 1 (15) | 1 (13) | 1 (1) | 4 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (3) | 5 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (6) | 1 (2) | 5 (6)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (5)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (3) | 1 (1) | 2 (2) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (6) | 2 (2) | 3 (6) | 8 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (6) | 1 (2) | 2 (2) | 6 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (5) | 2 (4) | 1 (2) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (3) | 1 (2) | 2 (2) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (2) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 2 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 1 (2) | 3 (4) | 6 (7)
Hypertension (Vascular disorders) | 1 (5) | 2 (12) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Jugular vein distension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02142049/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02142049/SAP_001.pdf